CLINICAL TRIAL: NCT03781388
Title: ED90 for Hyperbaric Bupivacaine in Spinal Anesthesia for Cesarean Delivery in Super Obese Parturients
Brief Title: ED90 for Hyperbaric Bupivacaine in Super Obese Parturients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00101530
Record Dates: First submitted 2018-12-18; First posted 2018-12-19 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Obesity, Morbid; Spinal Anesthesia; Cesarean Delivery
Keywords: Bupivacaine ED90; Cesarean Delivery; Obesity; Spinal Anesthesia
MeSH Terms: conditions — Obesity, Morbid; Obesity | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: The starting dose of hyperbaric bupivacaine for the first patient in this study will be 9mg; the dose for the subsequent subject will be based on the response of the preceding subject as per the Narayana Rule, a modification of the biased-coin design (BCD) up-down sequential method (UDM).
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Blinded study drugs will be prepared by an anesthesia provider not involved in the study. The anesthesia provider providing care to the patient will be blinded to the dosage of the hyperbaric bupivacaine. In order to preserve the blinding of the provider, the total volume of study drug will be maintained at a constant of 2.05mL. The difference in total volume based on the variation of hyperbaric bupivacaine dosing will be replaced with preservative free normal saline.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Starting dose of Bupivacaine (9 mg) (Experimental): The starting dose of hyperbaric bupivacaine for the first patient in this study will be 9mg; the dose for the subsequent subject will be based on the response of the preceding subject as per the Narayana Rule, a modification of the biased-coin design (BCD) up-down sequential method (UDM).
  Interventions: Drug: Bupivacaine
- Subsequent dose (Experimental)
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine — Determination of the dose will rely on the outcomes of the preceding 7 patients receiving the same dose, as the number of previous patients to consider is a function of the target dose. Among all patients who received a certain dose, a proportion of successful outcomes will be determined (P(d)); if P(d) <0.90, and at least one of the previous 7 patients who received the same dose had an unsatisfactory outcome, the next patient will receive a pre-determined increment of 0.75 mg of bupivacaine. Alternatively, if P(d) 0.90 and the previous 7 patients who received the same dose had successful outcomes, the next patient will receive a pre-determined decrement of 0.75mg of bupivacaine. Otherwise, the dose will remain the same.

SUMMARY:
The aim of this study is to determine the ED90 of hyperbaric intrathecal bupivacaine for the super obese population undergoing cesarean section under a combined spinal epidural technique.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology (ASA) class 2 and 3
* English speaking
* Gestational age > 36 weeks
* Scheduled for cesarean delivery under combined spinal epidural anesthesia
* 18 years or older
* BMI > 50 kg/m2

Exclusion Criteria:

* History of past or current intravenous drug or chronic opioid abuse
* Allergy or contraindication to any study medications
* Intrapartum cesarean delivery under epidural anesthesia
* Cesarean delivery under general anesthesia

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-12-06 (Actual); Study Completion 2022-12-06 (Actual)

PRIMARY OUTCOMES:
Percent of successful blocks for induction (success induction) | 10 minutes after intrathecal drug administration
  bilateral T6 sensory level to pinprick by
Percent of successful blocks for operation (success operation) | during surgery up to 90 minutes after intrathecal injection
  successful initial sensory level without requiring additional epidural anesthetic

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf S Habib, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tan HS, Fuller ME, Barney EZ, Diomede OI, Landreth RA, Pham T, Rubright SM, Ernst L, Habib AS. The 90% effective dose of intrathecal hyperbaric bupivacaine for Cesarean delivery under combined spinal-epidural anesthesia in parturients with super obesity: an up-down sequential allocation study. Can J Anaesth. 2024 May;71(5):570-578. doi: 10.1007/s12630-024-02705-5. Epub 2024 Mar 4. PMID 38438681